CLINICAL TRIAL: NCT06321276
Title: Investigation of the Efficiency of Radial Extracorporeal Shock Wave Therapy at Different Pulses in Patients With Carpal Tunnel Syndrom a Randomized Controlled Study
Brief Title: Investigation of the Efficiency of Radial Extracorporeal Shock Wave Therapy at Different Pulses in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Ibrahim Dogru, Physical medicine and rehabilitation MD, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEU-FTR-ID-01
Record Dates: First submitted 2024-01-03; First posted 2024-03-20 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: rehabilitation; extracorporeal shock wave therapy; physical therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: three groups with a conventional therapy control group
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- two thousand pulse ESWT Group (Active Comparator): ESWT will be applied to the patient's wrist and conventional treatment consisting of hand-wrist rest splint and nerve gliding exercises will be applied. The point of the ESWT site was located by ultrasonography interfaced with a 5-12 MHz linear array transducer, and the median nerve was visualized at the line of the proximal carpal tunnel (scaphoid pisiform level). (0,06 mj/mm2, 2000 impulses, 4 bar) (Modus ESWT Radial Shockwave Therapy)
  Interventions: Device: extracorporeal shockwave therapy
- one thousand pulse ESWT Group (Active Comparator): ESWT will be applied to the patient's wrist and conventional treatment consisting of hand-wrist rest splint and nerve gliding exercises will be applied. The point of the ESWT site was located by ultrasonography interfaced with a 5-12 MHz linear array transducer, and the median nerve was visualized at the line of the proximal carpal tunnel (scaphoid pisiform level). (0,06 mj/mm2, 1000 impulses, 4 bar) (Modus ESWT Radial Shockwave Therapy)
  Interventions: Device: extracorporeal shockwave therapy
- Conventional Control Group (No Intervention): The patient will receive conventional treatment consisting of hand-wrist rest splint and nerve gliding exercises as directed by the physiotherapist

INTERVENTIONS:
Device: extracorporeal shockwave therapy — Extracorporeal shock wave therapy (ESWT) is a non-invasive procedure that uses single-pulse acoustic waves generated outside the body and focused on a specific area of the body. Shock waves promote axonal regeneration of peripheral nerves through various molecular reactions. Although the anti-nociceptive mechanisms of ESWT have not yet been elucidated, ESWT may produce analgesia through biochemical changes in the nerve fiber itself and reduce inflammation of soft tissues.
  Arms: one thousand pulse ESWT Group; two thousand pulse ESWT Group

SUMMARY:
Different parameters have been used in studies investigating the efficacy of extracorporeal shock wave therapy in the treatment of carpal tunnel syndrome. Although extracorporeal shock wave therapy has been shown to have a positive effect on carpal tunnel syndrome, there is no consensus on which pulse rate is more effective. Therefore, in this study, the efficacy of extracorporeal shock wave therapy applied at different pulse rates in the treatment of carpal tunnel syndrome will be examined.

DETAILED DESCRIPTION:
The study included 72 patients with CTS aged 18-65 years who applied to Kırşehir Ahi Evran University Training and Research Hospital Physical Therapy and Rehabilitation Center.

Carpal tunnel syndrome (CTS) is the most common compressive neuropathy. In CTS, the median nerve is compressed within the carpal canal, about 1 to 2 cm beyond the distal wrist crease. It is more common in women and is typically more severe in the dominant hand but is often bilateral. Repetitive hand and wrist movements, such as using a keyboard or vibrating tools, have been associated with CTS. Medical conditions associated with CTS include diabetes, hypothyroidism and RA, as well as obesity and pregnancy. Rarely, CTS may be caused by a mass lesion in the wrist, such as a ganglion cyst or neurofibroma, or may be associated with acute trauma to the wrist. The vast majority of CTS cases are idiopathic.

CTS treatment is divided into conservative and surgical treatment. Conservative treatment methods are recommended in mild and moderate CTS patients, while surgical treatment is recommended in severe cases.

Extracorporeal Shock Wave Therapy is one of the physical therapy applications used in the treatment of Carpal Tunnel. The effectiveness of ESWT in the treatment of CTS will be examined

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-65 years with carpal tunnel syndrome diagnosed clinically and by EMG
* Patients who can correctly understand what is stated in the patient information form and who can cooperate
* Patients who consent to participate in the study according to the informed consent form will be included in the study.

Exclusion Criteria:

* Cervical radiculopathy
* Polyneuropathy
* Brachial plexopathy
* Use of systemic corticosteroids or local corticosteroid injections
* History of fracture and trauma in the forearm and wrist on the treated side
* Inflammatory rheumatic disease
* Pregnant and lactating patients
* Systemic diseases such as renal failure, peptic ulcer, DM, hypothyroidism, coagulation disorder
* Patients undergoing carpal tunnel syndrome surgery
* People with pacemakers
* Thoracic outlet syndrome
* Tenar atrophy, severe carpal tunnel syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 0. week , 4. week , 12. week
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity
Boston Carpal Tunnel Syndrome Questionnaire | 0. week, 4. week , 12. week
  It assesses the severity of symptoms and functional status. The symptom severity scale (SSS) assesses symptoms according to severity, frequency, time and type. The scale consists of 11 questions with multiple-choice answers scored from 1 point (mildest) to 5 points (most severe). The overall symptom severity score is calculated as the average of the scores for the 11 individual items.
  Functional status scale (FSS) assesses the impact of CTS on daily life. The scale consists of eight multiple-choice questions scored from 1 point (no difficulty in the activity) to 5 points (unable to do the activity at all). The total score for functional status was calculated as the average of all eight. Therefore, a higher symptom severity or functional status score indicates worse symptoms or impaired function.

SECONDARY OUTCOMES:
Hand grip strength measurement | 0. week, 4. week, 12. week
  Jamar hand dynamometer, which has high reliability and validity in many studies, will be used to measure hand grip strength. Hand grip strength will be measured in the recommended sitting position with the shoulder in adduction and neutral rotation, elbow in 90 degree flexion, forearm in midrotation and supported, and wrist in neutral. According to the test procedure, three consecutive measurements will be made for hand grip strength and the averages will be recorded in kg.
Electromyoneurography (EMNG) | 0. week, 12. week
  Median sensory nerve action potential amplitude, Compound muscle action potential amplitude, Median sensory distal latency, Median motor distal latency, Median sensory nerve conduction velocity, was evaluated by EMG.
Ultrasonography | 0. week, 12. week
  The cross-sectional area of the median nerve will be calculated by hand drawing with the existing program of the ultrasonography device. (The cross-sectional area, mm² ) The ratio of the length of the transverse diameter of the median nerve to the length of the longitudinal diameter will be used to obtain the flattening ratio (flattening ratio=FR, FR=the transverse diameter / the longitudinal diameter).

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim Doğru, MD, Principal Investigator — Kirsehir Ahi Evran University Physical medicine & rehabilitation
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huisstede BM, Hoogvliet P, Franke TP, Randsdorp MS, Koes BW. Carpal Tunnel Syndrome: Effectiveness of Physical Therapy and Electrophysical Modalities. An Updated Systematic Review of Randomized Controlled Trials. Arch Phys Med Rehabil. 2018 Aug;99(8):1623-1634.e23. doi: 10.1016/j.apmr.2017.08.482. Epub 2017 Sep 20. PMID 28942118
- [Background] Kim JC, Jung SH, Lee SU, Lee SY. Effect of extracorporeal shockwave therapy on carpal tunnel syndrome: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2019 Aug;98(33):e16870. doi: 10.1097/MD.0000000000016870. PMID 31415424
- [Background] Ozturk Durmaz H, Tuncay F, Durmaz H, Erdem HR. Comparison of Radial Extracorporeal Shock Wave Therapy and Local Corticosteroid Injection Effectiveness in Patients With Carpal Tunnel Syndrome: A Randomized Controlled Study. Am J Phys Med Rehabil. 2022 Jul 1;101(7):685-692. doi: 10.1097/PHM.0000000000001891. Epub 2021 Oct 4. PMID 35706121
- See also: Carpal Tunnel Syndrome: Effectiveness of Physical Therapy and Electrophysical Modalities. An Updated Systematic Review of Randomized Controlled Trials — https://pubmed.ncbi.nlm.nih.gov/28942118/
- See also: Effect of extracorporeal shockwave therapy on carpal tunnel syndrome: A systematic review and meta-analysis of randomized controlled trials — https://pubmed.ncbi.nlm.nih.gov/31415424/
- See also: Comparison of Radial Extracorporeal Shock Wave Therapy and Local Corticosteroid Injection Effectiveness in Patients With Carpal Tunnel Syndrome: A Randomized Controlled Study — https://pubmed.ncbi.nlm.nih.gov/35706121/